CLINICAL TRIAL: NCT06965621
Title: An Open-Label, Exploratory, Phase 2 Scintigraphy Study Evaluating 18F mFBG for Imaging Myocardial Sympathetic Innervation in Subjects With Heart Failure and Implantable Cardioverter-Defibrillators
Brief Title: 18F-mFBG Imaging for Myocardial Sympathetic Innervation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innervate Radiopharmaceuticals LLC (Formerly: Illumina Radiopharmaceuticals LLC) (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP101-221
Record Dates: First submitted 2025-03-20; First posted 2025-05-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy; ICD Patients
Keywords: Myocardial sympathetic innervation; PET myocardial imaging; 18F-mFBG
MeSH Terms: conditions — Heart Failure | interventions — Rubidium-82

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ischemic cardiomyopathy with ICD discharge (Active Comparator): 82Rb and 18F-mFBG will be administered to intraveously to 10 heart failure patients with ischemic cardiomyopathy and an ICD discharge within the past 12 months
  Interventions: Drug: 18F-metaFluorobenzylguanidine; Drug: Rubidium-82
- Ischemic cardiomyopathy without ICD discharge (Active Comparator): 82Rb and 18F-mFBG will be administered intravenously to 10 heart failure patients with ischemic cardiomyopathy and no ICD discharge within the past 12 months
  Interventions: Drug: 18F-metaFluorobenzylguanidine; Drug: Rubidium-82

INTERVENTIONS:
Drug: 18F-metaFluorobenzylguanidine — PET Radiopharmaceutical to assess myocardial sympathetic innervation
  Other Names: IRP101
Drug: Rubidium-82 — PET Radiopharmaceutical to assess myocardial perfusion

SUMMARY:
This is a Phase 2 study evaluating the positron-emitting radiopharmaceutical 18F-mFBG as an imaging agent for quantification of myocardial sympathetic innervation. The study will examine a group of stable patients with heart failure (HF) from ischemic cardiomyopathy. All subjects will have left ventricular ejection fraction (LVEF) ≤35% and implantable cardioverter-defibrillators (ICD). The primary objectives of the study will be to:

* document the degree to which 18F-mFBG uptake in the heart is reduced (compared to historical controls)
* characterize the distribution of regional abnormalities in relation to findings on rest/stress positron-emission tomography (PET) myocardial perfusion imaging (MPI)
* determine if there are global and/or regional differences in myocardial sympathetic innervation between subjects who have and have not experienced an appropriate ICD activation within the previous 12 months Effectiveness of 18F-mFBG will be judged in relation to historical experience with other nuclear imaging agents for cardiac sympathetic innervation imaging such as a 123I-meta-iodobenzylguanidine (mIBG) and 11C-hydroxyephedrine (HED).

Safety data will be collected to identify adverse events [AEs] and serious adverse events [SAEs] and characterize the safety profile of 18F-mFBG.

DETAILED DESCRIPTION:
The focus of most research into myocardial sympathetic neuronal imaging has been on NE analogues labeled with gamma- or positron-emitting radioisotopes. The most widely studied conventional nuclear imaging agent is 123I-metaiodobenzylguanidine (123I-mIBG), which provides effective and well-validated semi-quantitative information. In the pivotal trial (ADMIRE-HF) on which the US approval of 123I-mIBG for cardiac imaging was based, there was an increased occurrence of adverse outcomes (composite of HF progression, potentially fatal arrhythmias, and cardiac death) in HF subjects based upon the heart/mediastinum (H/M) ratio on late ("delayed") planar 123I-mIBG (AdreView™) images. Analyses of all-cause mortality in the ADMIRE-HFX extension study confirmed the low risk associated with H/M ≥1.60 (2-year mortality of 4%). Subsequent analyses specifically focused on arrhythmic events suggested that sympathetic neuronal imaging could aid in discriminating between low and higher risk cohorts. However, 123I-mIBG imaging results are heavily dependent on the imaging equipment and acquisition techniques used, and global standardization efforts have had limited success. In addition, absolute quantitation of myocardial uptake and clearance kinetics cannot be effectively achieved using single-photon emission computed tomography (SPECT), even with use of attenuation and scatter correction methods. These limitations and the high cost of the procedure have severely limited its use in clinical practice.

The preferred nuclear technique for high-resolution quantitative imaging of cellular functional behavior is PET. The present research will utilize a new 18F-labeled radiopharmaceutical, 18F-meta-fluorobenzylguanidine (18F-mFBG). The greatest advantage of this agent is its structural equivalence to 123I-mIBG, with the 123I atom in the latter replaced by a 18F atom.

The vast clinical and research experience with mIBG provides a strong basis for the expected performance of 18F-mFBG. In addition, animal and limited human experience suggests that clearance of 18F-mFBG from blood and certain target organs is more rapid than mIBG, such that target-background ratios (TBRs) for the heart should be superior for 18F-mFBG, improving both image quality and reliability of global and regional myocardial quantitation. To date, the focus of most research using 18F-mFBG has been on its use as an imaging agent for neural crest tumors such as neuroblastoma and pheochromocytoma (22). However, analyses of myocardial 18F-mFBG uptake in patients being evaluated for neural crest tumors suggested this agent could be effective as a cardiac imaging agent.

Past analyses of cardiac sympathetic imaging results have suggested this method might be of value for identifying heart disease patients at greater risk for arrhythmic events and sudden cardiac arrest (SCA). The largest prospective study on this topic enrolled 204 subjects eligible for implantable cardioverter defibrillators (LVEF ≤35%) who underwent cardiac PET imaging for myocardial sympathetic denervation using 11C-meta-hydroxyephedrine (11C-HED). The results showed that volume of denervated myocardium had the strongest correlation with SCA (arrhythmic death or defibrillator discharge). The 33 subjects with SCA had significantly larger denervated volumes than the 171 subjects without SCA (33±10% vs 26±11%; p<0.001). Multivariate analysis revealed that presence of 2 or more of risk factors of sympathetic denervation >37.6% of LV, LV end-diastolic index >99 ml/M2, creatinine >1.49 mg/dl, and no anti-angiotensin medication predicted a nearly 50% event rate over 4 years vs <1% annual rate without these risk factors (p < 0.0001).

The rationale for the present study is twofold.

1. Correlate areas of cardiac denervation with accurate measurements of regional cardiac blood flow (CBF) and inducible ischemia using standardized 82Rb PET.
2. Determine variables of sympathetic innervation and CBF most strongly related to past occurrence of arrhythmic events.

With the greater sensitivity and resolution of PET imaging compared to planar and SPECT techniques, it is expected that 18F -mFBG imaging will detect abnormalities that are missed with 123I mIBG and provide the reliable and reproducible quantitative accuracy necessary to support use of this agent for clinical patient studies.

ELIGIBILITY:
Inclusion Criteria:

* Stable heart failure from ischemic cardiomyopathy, LVEF < or = 35%, ICD implantation for at least 12 months

Exclusion Criteria:

* Unstable coronary artery disease, no ICD implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Quantify the degree of reduced myocardial 18F-mFBG uptake in adult HF subjects with well-characterized coronary heart disease | 24 hours from administration of the study drug for PET imaging and safety follow-up
  Obtain computer quantification of global and/or regional differences in myocardial sympathetic innervation (based on 18F-mFBG uptake) between subjects who have and have not experienced an appropriate ICD activation within the previous 12 months

SECONDARY OUTCOMES:
Quanify regional patterns of 18F-mFBG myocardial uptake and distribution | 24 hours from administration of the study drug for PET imaging and safety follow-up
  Obtain comparative computer quantification of regional patterns of 18F-mFBG myocardial uptake (sympathetic innervation) and areas of abnormal myocardial perfusion (blood flow) and/or wall motion (myocardial contraction) on PET myocardial perfusion imaging with Rubidium-82.
Perform Safety Data Collection for 18F-mFBG | 24 hours from administration of the study drug for safety follow-up
  Collect scheduled safety assessment data for 18F-mFBG Serious Adverse Events (SAE's) and Adverse Events (AE's).

CONTACTS AND LOCATIONS:
Overall Officials: K. Lance Gould, MD, Principal Investigator — Professor of Medicine, McGovern Medical School, UTHealth
Locations (1):
- UT Health Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a small Phase 2 study of an investigational drug; subject information will be available to the investigators and study sponsor only.

REFERENCES:
- [Background] Nakajima K, Verschure DO, Okuda K, Verberne HJ. Standardization of 123I-meta-iodobenzylguanidine myocardial sympathetic activity imaging: phantom calibration and clinical applications. Clin Transl Imaging. 2017;5(3):255-263. doi: 10.1007/s40336-017-0230-2. Epub 2017 May 4. PMID 28596948
- [Background] Verschure DO, Poel E, Travin MI, Henzlova MJ, Jain D, Jacobson AF, Verberne HJ. A simplified wall-based model for regional innervation/perfusion mismatch assessed by cardiac 123I-mIBG and rest 99mTc-tetrofosmin SPECT to predict arrhythmic events in ischaemic heart failure. Eur Heart J Cardiovasc Imaging. 2022 Aug 22;23(9):1201-1209. doi: 10.1093/ehjci/jeab132. PMID 34427293
- [Background] Travin MI, Henzlova MJ, van Eck-Smit BLF, Jain D, Carrio I, Folks RD, Garcia EV, Jacobson AF, Verberne HJ. Assessment of 123I-mIBG and 99mTc-tetrofosmin single-photon emission computed tomographic images for the prediction of arrhythmic events in patients with ischemic heart failure: Intermediate severity innervation defects are associated with higher arrhythmic risk. J Nucl Cardiol. 2017 Apr;24(2):377-391. doi: 10.1007/s12350-015-0336-8. Epub 2016 Jan 20. PMID 26791866
- [Background] Sood N, Al Badarin F, Parker M, Pullatt R, Jacobson AF, Bateman TM, Heller GV. Resting perfusion MPI-SPECT combined with cardiac 123I-mIBG sympathetic innervation imaging improves prediction of arrhythmic events in non-ischemic cardiomyopathy patients: sub-study from the ADMIRE-HF trial. J Nucl Cardiol. 2013 Oct;20(5):813-20. doi: 10.1007/s12350-013-9750-y. Epub 2013 Jul 18. PMID 23864400
- [Background] Narula J, Gerson M, Thomas GS, Cerqueira MD, Jacobson AF. (1)(2)(3)I-MIBG Imaging for Prediction of Mortality and Potentially Fatal Events in Heart Failure: The ADMIRE-HFX Study. J Nucl Med. 2015 Jul;56(7):1011-8. doi: 10.2967/jnumed.115.156406. Epub 2015 Jun 11. PMID 26069309
- [Background] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504